CLINICAL TRIAL: NCT03259230
Title: An Observational, Multicenter Study to Evaluate Interferon Gamma (IFNγ) and Other Inflammatory Mediators in Patients With Malignancy-Associated Hemophagocytic Lymphohistiocytosis (M-HLH)
Brief Title: Evaluation of IFNγ and Inflammatory Mediators in Patients With Malignancy-Associated Hemophagocytic Lymphohistiocytosis
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: NI-0501-07; PA16-0129 (Other: MD Anderson Cancer Center)
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Hemophagocytic Lymphohistiocytosis; Malignancy-Associated Hemophagocytic Lymphohistiocytosis; M-HLH; Patients with known diagnosis of malignancy without HLH; Interferon Gamma; IFNγ; Biomarkers; Inflammatory Markers; Blood draws; Data collection
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Approximate volume of 500 µl - 1 ml of serum or plasma required per time point. Minimum of 1 ml of whole blood collected for genetic characterization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malignancy-Associated Hemophagocytic Lymphohistiocytosis: Patients diagnosed with HLH in the context of a malignancy. The diagnosis of M-HLH was established by the treating physician.
  Interventions: Other: Blood Draws; Other: Data Collection
- Absence of HLH in patients diagnosed with malignancy: Patients with a diagnosis of hematological malignancy and never diagnosed with HLH or no suspicion of HLH (at any time, including time after sample collection in case of use of retrospective sample).
  Interventions: Other: Blood Draws; Other: Data Collection

INTERVENTIONS:
Other: Blood Draws
Other: Data Collection

SUMMARY:
This observational study is designed to determine the levels of pro-inflammatory markers in patients diagnosed with M-HLH, and to assess whether the cytokine profiles bear an IFNγ signature.

DETAILED DESCRIPTION:
This is a observational study designed to determine the levels of inflammatory markers in patients diagnosed with M-HLH and to assess the relationship between the biomarkers and disease activity in these patients during the M-HLH course. Inflammatory markers will also be measured in a group of control patients diagnosed with hematological malignancy but without HLH. Inflammatory markers include IFNγ and IFNγ-induced chemokines CXCL9 and CXCL10.

In addition to the blood samples for the biomarker analysis, relevant information gathered by the treating physician will be collected in a data collection form. Whenever possible, collection of serum samples for biomarker analysis and relevant information should occur at M-HLH diagnosis, at regular time intervals during the treatment course as well as at resolution or reactivation of the disease.

Blood samples will also be sent to the study sponsor (NovImmune S.A.) for cytokine testing. Before participant's samples are sent to the sponsor for testing, participant's name and any personal identifying information will be coded to protect participant's privacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with HLH in the context of a malignancy. The diagnosis of M-HLH will be established by the treating physician.
2. The patient or patient's legal representative (in case the patient is < 18 years old) must have consented to the use of their clinical data for research purposes at the site.
3. For the control group, patients with a diagnosis of hematological malignancy and never diagnosed with HLH or no suspicion of HLH

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female (adult and children) patients who are diagnosed with M-HLH and that meet the inclusion criteria. In addition, patients with a diagnosis of hematological malignancy in the absence of HLH will be included as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 4 observational study was conducted in patients diagnosed with malignancy-associated hemophagocytic lymphohistiocytosis (M-HLH) at a single center in the United States of America.
Pre-assignment Details: A total of 40 patients were enrolled in the study. Of which 39 patients had a confirmed malignancy and were included in the malignancy set for analysis.
Groups:
- Hemophagocytic Lymphohistiocytosis (HLH) Patients: All patients diagnosed with HLH in the context of a malignancy.
- Non-HLH Patients: All patients with a diagnosis of hematological malignancy and never diagnosed with HLH or no suspicion of HLH (at any time, including time after sample collection in case of use of retrospective sample).
Period: Overall Study
Arm/Group | Hemophagocytic Lymphohistiocytosis (HLH) Patients | Non-HLH Patients
Started | 20 | 20
Malignancy Analysis Set | 19 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Excluded from the Malignancy Analysis Set | 1 | 0

BASELINE CHARACTERISTICS:
Population: The malignancy set included all patients who were diagnosed with malignancy.
Groups:
- HLH Patients: All patients diagnosed with HLH in the context of a malignancy.
- Total: Total of all reporting groups
Arm/Group | HLH Patients | Non-HLH Patients | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (18.6) | 63.2 (15.3) | 60.0 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 15 | 12 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - C-X-C Chemokine Ligand 10 (CXCL10)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of CXCL10.
Time Frame: From Day 1 up to 39.5 months
Population: The malignancy set included all patients who were diagnosed with malignancy. Only patients with data available are reported.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 19 | 5
picogram/milliliter (pg/mL) | 5040.638 (9622.745) | 454.392 (246.307)

2. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - C-X-C Chemokine Ligand 9 (CXCL9)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of CXCL9.
Time Frame: From Day 1 up to 39.5 months
Population: The malignancy set included all patients who were diagnosed with malignancy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 19 | 19
pg/mL | 8878.698 (17582.571) | 1864.255 (4986.931)

3. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Interferon Gamma (IFNg)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of IFNg.
Time Frame: From Day 1 up to 39.5 months
Population: The malignancy set included all patients who were diagnosed with malignancy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 19 | 19
pg/mL | 279.951 (898.740) | 8.014 (2.370)

4. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Interleukin 10 (IL-10)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of IL-10.
Time Frame: From Day 1 up to 39.5 months
Population: The malignancy set included all patients who were diagnosed with malignancy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 19 | 19
pg/mL | 46.562 (124.537) | 2.185 (2.953)

5. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Interleukin 1 Beta (IL-1B)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of IL-1B.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 19 | 5
pg/mL | 2.140 (0.000) | 2.140 (0.000)

6. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Interleukin 6 (IL-6)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of IL-6.
Time Frame: From Day 1 up to 39.5 months
Population: The malignancy set included all patients who were diagnosed with malignancy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 19 | 19
pg/mL | 597.385 (1776.853) | 10.059 (28.771)

7. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Neopterin
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of neopterin.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanomoles
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 14 | 19
nanomoles | 257.120 (223.475) | 51.909 (47.869)

8. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Tumor Necrosis Factor Alpha (TNFa)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of TNFa.
Time Frame: From Day 1 up to 39.5 months
Population: The malignancy set included all patients who were diagnosed with malignancy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 19 | 19
pg/mL | 12.412 (14.899) | 4.751 (4.054)

9. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Total Human Interferon Gamma (hIFNg)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of hIFNg.
Time Frame: From Day 1 up to 39.5 months
Population: The malignancy set included all patients who were diagnosed with malignancy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 19 | 19
pg/mL | 82.227 (196.240) | 417.603 (1573.368)

10. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Soluble CD163 (sCD163)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of sCD163.
Time Frame: From Day 1 up to 39.5 months
Population: The malignancy set included all patients who were diagnosed with malignancy.
Measure: Mean (Standard Deviation); unit: nanogram/mL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 19 | 19
nanogram/mL | 3796.175 (3154.561) | 1812.384 (2852.523)

11. Primary Outcome: Mean Serum Concentration of Inflammatory Biomarker - Soluble IL-2 Receptor Alpha (sIL2Ra)
Description: Serum samples was collected at various times after HLH diagnosis to determine the concentration of sIL2Ra.
Time Frame: From Day 1 up to 39.5 months
Population: The malignancy set included all patients who were diagnosed with malignancy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 19 | 19
pg/mL | 10183.509 (12244.564) | 2575.569 (3395.536)

12. Primary Outcome: Mean Serum Concentration of Hemoglobin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of hemoglobin.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gram/deciliter (g/dL)
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
gram/deciliter (g/dL) | 9.31 (0.98) | 8.52 (1.95)

13. Primary Outcome: Mean Serum Concentration of Hematocrit
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of hematocrit.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter (L) of cells/L of blood
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
liter (L) of cells/L of blood | 27.28 (3.41) | 25.94 (4.99)

14. Primary Outcome: Mean Serum Concentration of Erythrocytes
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of erythrocytes.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^12/L
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
cells*10^12/L | 3.208 (0.371) | 2.896 (0.543)

15. Primary Outcome: Mean Serum Concentration of Leukocytes
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of leukocytes.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
cells*10^9/L | 2.11 (2.85) | 8.42 (8.94)

16. Primary Outcome: Mean Serum Concentration of Neutrophils
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of neutrophils.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^3/microliter (mcL)
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
cells*10^3/microliter (mcL) | 1.743 (2.550) | 1.984 (1.776)

17. Primary Outcome: Mean Serum Concentration of Lymphocytes
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of lymphocytes.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
cells*10^3/mcL | 0.468 (0.647) | 0.968 (1.084)

18. Primary Outcome: Mean Serum Concentration of Monocytes
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of monocytes.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 10 | 5
cells*10^3/mcL | 0.233 (0.272) | 1.278 (1.034)

19. Primary Outcome: Mean Serum Concentration of Eosinophils
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of eosinophils.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 4 | 3
cells*10^3/mcL | 0.032 (0.044) | 1.083 (1.441)

20. Primary Outcome: Mean Serum Concentration of Basophils
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of basophils.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 2 | 2
cells*10^3/mcL | 0.100 (0.087) | 0.820 (0.834)

21. Primary Outcome: Mean Serum Concentration of Platelets
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of platelets.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*10^3/mcL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
cells*10^3/mcL | 43.9 (67.7) | 30.8 (38.5)

22. Primary Outcome: Mean Plasma Concentration of Fibrinogen
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of fibrinogen.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram (mg)/dL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 2
milligram (mg)/dL | 207.5 (143.0) | 357.5 (2.1)

23. Primary Outcome: Mean Plasma Concentration of D-Dimer
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of D-dimer.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram (mcg)/mL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 15 | 2
microgram (mcg)/mL | 10.165 (7.569) | 2.220 (2.107)

24. Primary Outcome: Mean Serum Concentration of Ferritin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of ferritin.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 2
mcg/L | 17240.3470 (30134.8903) | 3.8940 (4.1748)

25. Primary Outcome: Mean Serum Concentration of Fasting Triglycerides
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of fasting triglycerides.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 16 | 0
mg/dL | 231.5 (88.6) |

26. Primary Outcome: Mean Serum Concentration of Creatinine
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of creatinine.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 4
mg/dL | 1.682 (2.726) | 0.808 (0.287)

27. Primary Outcome: Mean Plasma Concentration of Blood Urea Nitrogen
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of blood urea nitrogen.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 13 | 4
mg/dL | 44.68 (30.53) | 29.00 (3.92)

28. Primary Outcome: Mean Serum Concentration of Albumin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of albumin.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 4
g/dL | 2.88 (0.60) | 3.48 (0.82)

29. Primary Outcome: Mean Serum Concentration of Sodium
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of sodium.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimoles/L
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 4
millimoles/L | 137.3 (7.4) | 139.5 (4.1)

30. Primary Outcome: Mean Serum Concentration of Beta2-Microglobulin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of beta2-microglobulin.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 10 | 1
mg/L | 9.48 (15.19) | 3.10 (NA) — Standard deviation is not applicable for N=1.

31. Primary Outcome: Mean Serum Concentration of Immunoglobulin G (IgG)
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of IgG.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 15 | 2
mg/dL | 602.2 (250.6) | 722.0 (353.6)

32. Primary Outcome: Mean Serum Concentration of C-Reactive Protein
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of c-reactive protein.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 13 | 0
mg/dL | 102.508 (174.824) |

33. Primary Outcome: Mean Serum Concentration of Aspartate Aminotransferase
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of aspartate aminotransferase.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: international units/L (IU/L)
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 17 | 4
international units/L (IU/L) | 177.8 (279.9) | 44.8 (18.4)

34. Primary Outcome: Mean Serum Concentration of Alanine Aminotransferase
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of alanine aminotransferase.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
IU/L | 127.9 (179.0) | 34.0 (25.4)

35. Primary Outcome: Mean Serum Concentration of Alkaline Phosphatase
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of alkaline phosphatase.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
IU/L | 216.0 (170.5) | 95.0 (74.5)

36. Primary Outcome: Mean Serum Concentration of Lactate Dehydrogenase
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of lactate dehydrogenase.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
IU/L | 7469.5 (10456.7) | 1100.8 (718.5)

37. Primary Outcome: Mean Serum Concentration of Total Bilirubin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of total bilirubin.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 18 | 5
mg/dL | 2.64 (3.85) | 1.68 (1.40)

38. Primary Outcome: Mean Serum Concentration of Conjugated Bilirubin
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of conjugated bilirubin.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 15 | 1
mg/dL | 1.96 (3.71) | 0.00 (NA) — Standard deviation is not applicable for N=1.

39. Primary Outcome: Mean Serum Concentration of Natural Killer (NK) Cell Activity
Description: Blood samples was collected at various times after HLH diagnosis to determine the concentration of NK cell activity. A lytic unit 30 (LU30) was defined as the number of effector cells necessary to cause lysis of 30% of its target cells.
Time Frame: From Day 1 up to 39.5 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: LU30
Arm/Group | HLH Patients | Non-HLH Patients
Number analyzed (Participants) | 2 | 0
LU30 | 3.5 (0.7) |

ADVERSE EVENTS:
Description: Safety analysis including all-cause mortality, serious adverse events and other (non-serious) adverse events were not monitored as this is an observational study.
Arm/Group | HLH Patients | Non-HLH Patients
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT03259230/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT03259230/SAP_001.pdf